CLINICAL TRIAL: NCT05607277
Title: Global Iliac Branch Study (Iliac Conformability Paper, Gore vs. Cook)
Brief Title: Global Iliac Branch Study
Acronym: GIBS
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0677; A539750 (Other: UW Madison); SMPH/SURGERY/VASCULAR SURGERY (Other: UW Madison); Protocol Version 7/29/2020 (Other: UW Madison)
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2022-10

CONDITIONS: Abdominal Aortic Aneurysm; Iliac Aneurysm
Keywords: Abdominal aortic aneurysm; Aorta-Iliac aneurysm; Endovascular aneurysm repair; Iliac Branch Devices
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Procedure: Endovascular Repair of abdominal aortic aneurysms — Femoral artery access
  Other Names: Endovascular repair of abdominal aorto-iliac aneurysm

SUMMARY:
This project seeks to determine if certain anatomic factors, specifically tortuous and non-conformable iliac arteries, may predict device complications, including seal zone failure, type III endoleak, and occlusion. Approximately 400 subjects from 5 academic centers across the United States, Europe, and Asia will be included in this study. Various markers of pre- and post-treatment iliac anatomy will be measured using CT imaging, and clinical events will be reported by academic centers. The relationship of imaging data to patient demographics will then be assessed alongside anatomic and demographic predictors of non-conformability.

DETAILED DESCRIPTION:
Background and significance Abdominal aortic aneurysms (AAAs) affect 0.5% to 1.3% of women and 4.0% to 7.6% of men age 65 and older1-4. Infrarenal AAAs frequently extend distally through the aortic bifurcation and into the common, external, and/or internal iliac arteries,5,6 presenting a challenge for aneurysm repair. Current guidelines prioritize repair strategies which preserve blood flow to the internal iliac artery (IIA) with the goal of reducing the complications of buttock claudication and pelvic ischemia.7-9 As endovascular intervention has become standard practice for those with eligible anatomy, 7 branched endovascular devices have been developed to preserve IIA blood flow when repairing AAAs with iliac involvement.

With the ongoing development of devices and techniques, the range of iliac anatomy eligible for endovascular repair has increased. Most notably, multiple iliac branch devices (IBDs) are being used to treat AAAs involving highly tortuous iliac arteries. A variety of IBDs are available globally, and as such, there is an opportunity to determine if certain anatomic factors- specifically tortuous and non-conformable iliac arteries- may predict device complications.

To begin exploring this question, the Global Iliac Branch Study (GIBS)- a partnership between 5 centers across the United States, Europe, and Asia- was developed to evaluate performance of branched endografts based on anatomical assessments, with analysis of CT scans using centralized and standardized analysis protocols at the AortaCore Imaging Lab at the University of Wisconsin-Madison.

Previous work In addition to elevated risk of conversion to open repair,10 iliac tortuosity has previously been associated with increased risk of "conformability" events, including seal zone failure, type III endoleak, occlusion, stenosis, compression, and device migration.11-13

Previously, the applicant and her faculty mentor have explored the interaction between iliac tortuosity and device conformability in patients treated with the W.L.GORE EXCLUDER iliac branch endoprosthesis (IBE).14 Non-conformation was defined as a decrease in the total iliac index of tortuosity beyond 15%. This study found that non-conformation, as well as internal iliac artery diameter of less than 10 mm, were associated with adverse iliac events after iliac branch endoprosthesis (odds ratio, 8.2 [P = .02] and odds ratio, 12.3 [P = .02], respectively).

Similar to the aforementioned studies demonstrating increasing ranges of anatomic eligibility with the development of more complex and accommodating devices, the applicant and her mentor explored device eligibility for endovascular repair (EVAR) of small AAA over two years in a paper published in November 2021 in the Journal of Vascular Surgery which found high levels of anatomic eligibility for EVAR at baseline, and preservation of this eligibility over two years.15 These findings, like those previously mentioned, suggested that advancements in EVAR device design have improved anatomic eligibility for the procedure. Compared to open repair, EVAR is associated with decreased periprocedural morbidity and hospital length of stay,16 and as such is the preferred approach, as well as a major target for innovation in the field of vascular surgery.

Methods and analysis CT images of 400 subjects with IBDs from 5 centers around the globe will be transferred and analyzed at the University of Wisconsin-Madison AortaCore Imaging Lab under an Institutional Review Board (IRB) approved protocol. Post-processing workstations using Aquarius Intuition (version 4.4.12, TeraRecon) will be used to measure morphology data. Each CT will be fit with a manually corrected centerline that is equidistant from the outer walls of the aneurysmal vessels. Measurements will be completed at both the pre-treatment and post-treatment intervals; these include common, external, and internal iliac artery diameters and lengths, common iliac artery index of tortuosity (Common Iliac Index; Centerline length of the common iliac artery (CIA) divided by the shortest straight-line distance between the CIA origin and iliac bifurcation), total iliac artery index of tortuosity (Total Iliac Index; centerline length of the CIA plus centerline length of the external iliac artery, divided by the shortest straight-line distance between the CIA origin and terminal external iliac artery), and presence of the double iliac sign (when any portion of the iliac vessel is tortuous enough to be duplicated in a single cut of an axial computed tomography slice.)17 Figures 1 and 2 demonstrate these measurement techniques for capturing and quantifying tortuosity.

Measurement of these values before and after device deployment allows the determination of differences in iliac artery length pre- and post-treatment, which is used to quantify device "conformability."18 Notably, devices which produce minimal changes to native anatomy are considered more "conformable" and devices that make greater changes to iliac lengths and angle anatomy are considered "non-conformable" (Figure 3.)

In addition to pre-treatment demographics and comorbidities, including age, sex, and geographic origin, associations between iliac tortuosity indices and the aforementioned CT measurements will be determined in relation to clinical events collected by each center including conversion to open repair, re-intervention, endoleak, occlusion, compression, patient-reported symptoms and adverse events, and death.

Continuous variables will be compared using the unpaired Student t test if normally distributed and the Mann-Whitney U test or Wilcoxon matched pairs test if they are not normally distributed. Categorical variables will be compared using the Fisher exact test or Pearson's x2 test.

Expected outcomes As previously described, in preliminary data14 we have identified that a postoperative change in iliac tortuosity ("non-conformability") predicts adverse events in a sample size of 98 patients. We hypothesize that a larger sample size of 400 patients will confirm this relationship between non-conformability and adverse events, and enable identification of pre-operative predictors of non-conformability. Furthermore, we anticipate that the inclusion of a more diverse selection of endovascular devices will more broadly capture the relationship between device conformability and iliac tortuosity beyond what can be determined based on commercially available devices in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone endovascular aortic repair of AAA with iliac involvement via iliac branch device.

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 subjects with Endovascular repair with Iliac Branched Devices for treatment of abdominal aortic aneurysm with iliac involvement.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Device conformability in relation to endovascular repair of abdominal aortoiliac aneurysms. | Pre-treatment
  Adverse events: any radiographic or clinical ipsilateral complication, i.e. dissection, kink, compression, occlusion, endoleaks.
Device conformability in relation to endovascular repair of abdominal aortoiliac aneurysms. | 1 day at First post-operative imaging appointment
  Adverse events: any radiographic or clinical ipsilateral complication, i.e. dissection, kink, compression, occlusion, endoleaks.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Matsumura, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chichester Aneurysm Screening Group; Viborg Aneurysm Screening Study; Western Australian Abdominal Aortic Aneurysm Program; Multicentre Aneurysm Screening Study. A comparative study of the prevalence of abdominal aortic aneurysms in the United Kingdom, Denmark, and Australia. J Med Screen. 2001;8(1):46-50. doi: 10.1136/jms.8.1.46. PMID 11373850
- [Background] Derubertis BG, Trocciola SM, Ryer EJ, Pieracci FM, McKinsey JF, Faries PL, Kent KC. Abdominal aortic aneurysm in women: prevalence, risk factors, and implications for screening. J Vasc Surg. 2007 Oct;46(4):630-635. doi: 10.1016/j.jvs.2007.06.024. PMID 17903646
- [Background] US Preventive Services Task Force; Owens DK, Davidson KW, Krist AH, Barry MJ, Cabana M, Caughey AB, Doubeni CA, Epling JW Jr, Kubik M, Landefeld CS, Mangione CM, Pbert L, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Abdominal Aortic Aneurysm: US Preventive Services Task Force Recommendation Statement. JAMA. 2019 Dec 10;322(22):2211-2218. doi: 10.1001/jama.2019.18928. PMID 31821437
- [Background] Svensjo S, Bjorck M, Wanhainen A. Current prevalence of abdominal aortic aneurysm in 70-year-old women. Br J Surg. 2013 Feb;100(3):367-72. doi: 10.1002/bjs.8984. Epub 2012 Nov 28. PMID 23192439
- [Background] Ghosh J, Murray D, Paravastu S, Farquharson F, Walker MG, Serracino-Inglott F. Contemporary management of aorto-iliac aneurysms in the endovascular era. Eur J Vasc Endovasc Surg. 2009 Feb;37(2):182-8. doi: 10.1016/j.ejvs.2008.11.001. Epub 2008 Nov 29. PMID 19046903
- [Background] Maurel B, Bartoli MA, Jean-Baptiste E, Reix T, Cardon A, Goueffic Y, Martinez R, Cochennec F, Albertini JN, Chauffour X, Steinmetz E, Haulon S; Association Universitaire de Recherche en Chirurgie Vasculaire, France. Perioperative evaluation of iliac ZBIS branch devices: a French multicenter study. Ann Vasc Surg. 2013 Feb;27(2):131-8. doi: 10.1016/j.avsg.2011.02.052. PMID 23380549
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Faries PL, Morrissey N, Burks JA, Gravereaux E, Kerstein MD, Teodorescu VJ, Hollier LH, Marin ML. Internal iliac artery revascularization as an adjunct to endovascular repair of aortoiliac aneurysms. J Vasc Surg. 2001 Nov;34(5):892-9. doi: 10.1067/mva.2001.118085. PMID 11700492
- [Background] Kouvelos GN, Katsargyris A, Antoniou GA, Oikonomou K, Verhoeven EL. Outcome after Interruption or Preservation of Internal Iliac Artery Flow During Endovascular Repair of Abdominal Aorto-iliac Aneurysms. Eur J Vasc Endovasc Surg. 2016 Nov;52(5):621-634. doi: 10.1016/j.ejvs.2016.07.081. Epub 2016 Sep 2. PMID 27600731
- [Background] Cuypers PW, Laheij RJ, Buth J. Which factors increase the risk of conversion to open surgery following endovascular abdominal aortic aneurysm repair? The EUROSTAR collaborators. Eur J Vasc Endovasc Surg. 2000 Aug;20(2):183-9. doi: 10.1053/ejvs.2000.1167. PMID 10944101
- [Background] Iwakoshi S, Nakai T, Ichihashi S, Inoue T, Sakaguchi S, Hirose T, Tabayashi N, Watkins AC, Kichikawa K. Conformability and Efficacy of the Zenith Spiral Z Leg Compared with the Zenith Flex Leg in Endovascular Abdominal Aortic Aneurysm Repair. Ann Vasc Surg. 2019 Aug;59:127-133. doi: 10.1016/j.avsg.2019.02.013. Epub 2019 May 7. PMID 31071429
- [Background] Wolf YG, Tillich M, Lee WA, Rubin GD, Fogarty TJ, Zarins CK. Impact of aortoiliac tortuosity on endovascular repair of abdominal aortic aneurysms: evaluation of 3D computer-based assessment. J Vasc Surg. 2001 Oct;34(4):594-9. doi: 10.1067/mva.2001.118586. PMID 11668310
- [Background] Parra JR, Ayerdi J, McLafferty R, Gruneiro L, Ramsey D, Solis M, Hodgson K. Conformational changes associated with proximal seal zone failure in abdominal aortic endografts. J Vasc Surg. 2003 Jan;37(1):106-11. doi: 10.1067/mva.2002.53. PMID 12514585
- [Background] DeRoo E, Harris D, Olson S, Panthofer A, Meadows W, Pauli T, Peterson B, Schneider D, Matsumura J. Conformability of the GORE EXCLUDER iliac branch endoprosthesis is associated with freedom from adverse iliac events. J Vasc Surg. 2021 Nov;74(5):1558-1564.e1. doi: 10.1016/j.jvs.2021.05.026. Epub 2021 Jun 1. PMID 34082005
- [Background] Panthofer AM, Olson SL, Rademacher BL, Grudzinski JK, Chaikof EL, Matsumura JS; N-TA(3)CT Investigators. Anatomic eligibility for endovascular aneurysm repair preserved over 2 years of surveillance. J Vasc Surg. 2021 Nov;74(5):1527-1536.e1. doi: 10.1016/j.jvs.2021.04.044. Epub 2021 May 4. PMID 33957227
- [Background] Olson SL, Panthofer AM, Harris DJ, Jordan WD Jr, Farber MA, Cambria RP, Matsumura JS. CT-Derived Pretreatment Thoracic Sarcopenia Is Associated with Late Mortality after Thoracic Endovascular Aortic Repair. Ann Vasc Surg. 2020 Jul;66:171-178. doi: 10.1016/j.avsg.2019.10.089. Epub 2019 Nov 6. PMID 31705993